CLINICAL TRIAL: NCT05078983
Title: Investigation of Relation With Preoperative Fragility and ASA Score in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sultan Keskin Demircan, Principal Investigator, Gulhane Training and Research Hospital
Other Study IDs: 2021/11
Record Dates: First submitted 2021-09-22; First posted 2021-10-15 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Frail Elderly Syndrome; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIGH RISK: HIGH RISK MEANS PATIENTS HAVE ASA SCORE OVER 2
  Interventions: Diagnostic Test: CGA-FI (COMPREHENSIVE GERIATRIC ASSESMENT - FRAILITY INDEX)
- LOW RISK: LOW RISK MEANS PATIENTS HAVE ASA SCORE BELOW 3
  Interventions: Diagnostic Test: CGA-FI (COMPREHENSIVE GERIATRIC ASSESMENT - FRAILITY INDEX)

INTERVENTIONS:
Diagnostic Test: CGA-FI (COMPREHENSIVE GERIATRIC ASSESMENT - FRAILITY INDEX) — GERIATRIC ASSESMENT TEST

SUMMARY:
Frailty is a term specific to the geriatric period. It is used to describe weak, unstable, frail patients and partially expresses the frailty of the elderly patient. Once the frailty process begins, the risk of loss of mobility, dependency and mortality increases.

Frailty is an important predictor of adverse outcomes after surgery. According to studies conducted in various surgical situations, fragility is a major risk factor for morbidity, mortality and longer hospital stay. According to the available data, frailty has a sufficient basis for determining the risks of patients before surgery, developing preventive methods and making personal treatment decisions. As the frailty index increased, it was observed that the duration of postoperative hospital stay was associated with the need for intensive care, postoperative complications, and the rate of re-admissions within 30 days.

ASA (American Society of Anesthesiologists) classification is widely used in order to evaluate the physical condition preoperatively in geriatric individuals with multiple comorbidities. Considering the fragility variable while creating the ASA score in the preoperative period may be useful in determining the follow-up strategy during the operation and postoperative period. For example, a patient who is evaluated as ASA 2 because he has no problems other than simple 1-2 comorbid conditions, involuntary weakening of 5% in the last 1 year (not easily noticed), weakness (can only be detected with a dynamometer) and cessation of going out of the house (can only be understood when asked privately). ) can be categorized as at risk at ASA level 3-4, as it is understood to be fragile.

The aim of this project is to examine the frequency of frailty in elderly individuals who will be operated on, and to examine the relationship between frailty and ASA score using the anthropometry and comorbidity differences between frail preoperative patients and those who do not.

ELIGIBILITY:
Inclusion Criteria:

- Patients over the age of 65 who were admitted to the general surgery service for surgery and then operated.

Exclusion Criteria:

-Patients with advanced stage dementia

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients over the age of 65 who were admitted to the general surgery service for surgery and then operated.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-10-17 (Estimated); Study Completion 2022-11-17 (Estimated)

PRIMARY OUTCOMES:
DEATH RATE | AT 1 MONTH AND 3 MONTH AFTER OPERATION
  PROPORTION OF PATIENTS WHO DIED TO ALL PATIENTS
LENGTH OF HOSPITAL STAY | AT 1 MONTH
  NUMBER OF NIGHTS THE PATIENT NEEDS TO STAY IN HOSPITAL
DELIRIUM RATE | AT 1 MONTH
  THE RATIO OF THE NUMBER OF PATIENTS IN DELIRIUM TO THE TOTAL NUMBER OF PATIENTS AFTER OPERATION
INTENSIVE CARE RATE | AT 1 MONTH
  THE RATIO OF THE NUMBER OF PATIENTS NEED INTENSIVE CARE AFTER OPERATION TO TOTAL NUMBER OF PATIENTS

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane training and research hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided